CLINICAL TRIAL: NCT03105674
Title: Multi-drug Analgesia Versus Standard Solution for Perianal Block - A Prospective Study to Determine the Efficacy, Cost and Narcotic Consumption in the Post-operative Period
Brief Title: Multi-Drug Analgesia vs. Standard Solution for Anal Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Not yet IRB approved and PI will be leaving institution in September.
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AAAQ9398
Record Dates: First submitted 2017-03-16; First posted 2017-04-10 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Hemorrhoids; Fissure in Ano; Fistula;Rectal
Keywords: analgesia; peri-anal procedure; peri-anal block; anal surgery
MeSH Terms: conditions — Hemorrhoids; Fissure in Ano; Rectal Fistula; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard Therapy (Active Comparator): Patients will receive a combination of Marcaine and Lidocaine injection (standard local anesthetics) as a part of their peri-anal block prior to the surgery.
  Interventions: Drug: Standard local anesthetics (Combination)
- Multi-drug local anaesthetics (Experimental): Patients will receive a combination [Multi-drug local anesthetics (Combination)] of following drugs as a part of their peri-anal block prior to the surgery (multi-drug local anesthetics)
  1. Ropivacaine 0.5% - 30 ml
  2. Ketorolac 30mg/ml - 1 ml
  3. Kenalog 10 mg/ml - 5 ml
  4. Lidocaine 1% with Epinephrine 1:100,000 - 20ml
  Interventions: Drug: Multi-drug local anesthetics (Combination)

INTERVENTIONS:
Drug: Multi-drug local anesthetics (Combination) — 1. Ropivacaine 0.5% - 30 ml
  2. Ketorolac 30mg/ml - 1 ml
  3. Kenalog 10 mg/ml - 5 ml
  4. Lidocaine 1% with Epinephrine 1:100,000 - 20ml
  Other Names: Peri-anal block
  Arms: Multi-drug local anaesthetics
Drug: Standard local anesthetics (Combination) — Marcaine and Lidocaine
  Other Names: Standard solution
  Arms: Standard Therapy

SUMMARY:
The primary aim is to test the magnitude and duration of analgesia provided by single dose multi-drug analgesia administered for perianal block, and compare with standard solution (Marcaine & Lidocaine in 1:1 mixture - Total 60 ml), at post-operative period and also to compare with the standard solution including their respective post-operative opioid or non-opioid oral analgesic requirement. Local anesthesia via a perianal block using multi-drug analgesia or standard solution will be compared using the Numeric pain rating scale on Post-operative day 1, 3 and during follow up visit on day 7. The investigators hope to find a better control of post-operative analgesia which will lead to better functional outcomes. Possible decrease consumption of opioids in the post-operative period will perhaps decrease the cost and chances of addiction and will increase patient comfort and compliance.

DETAILED DESCRIPTION:
Post-operative analgesia after anorectal surgery still poses a significant problem. Technical or operator dependent factors have been proposed for causing severe pain post operatively. Many factors such as height of anastomosis, incorporation of smooth muscle, size of doughnut, and inclusion of squamous epithelium were considered to cause pain specially after hemorrhoidectomy. However, in spite of standardizing the techniques, patients still experience moderate to severe pain after anorectal surgery. Effective post-surgical pain control is critical to patient recovery, and can contribute to improved healing, faster patient mobilization, reduced hospital stays and health care costs. Effective multimodal techniques have been devised to maximize pain relief, lower the risk of adverse events, and improve patient outcomes. These techniques (wound infiltration with local anesthetic being most common) is short lived, maximum up to 12 hours. Post-operative pain usually lasts for 72 hours and thus the systemic opioids remain the mainstay pain control post-operatively. Although effective analgesics, they are associated with unwanted and potentially adverse events, such as nausea, vomiting, pruritus, sedation, cognitive impairment, urinary retention, sleep disturbances, and respiratory depression. Also, narcotic addiction remains a concern for surgical patients. Some patients would like to have effective analgesia and thus also avoid narcotics.Multi-drug analgesic combinations are used in orthopedic surgery (Ropivacaine, Ketorolac, and Morphine, with adrenaline) and during hemorrhoidectomy (extended-release liposome Bupivacaine) which showed decrease in post-operative analgesia requirement. However, no studies that used multi-drug analgesia show any effect on the pain medication consumption after discharge for ambulatory surgery. The investigators have designed a novel multi-drug anesthetic formulation to achieve long-acting postoperative analgesia with single-dose administration intra-operative via perianal block and wound infiltration.

ELIGIBILITY:
Inclusion Criteria:

* Men and nonpregnant women aged 18 years or older scheduled to undergo anorectal procedures
* Female patients must be postmenopausal, surgically sterile, or willing to use acceptable means of contraception for at least 30 days after surgery.
* Patients will be required to have an Americal society of anesthesia physical status classification of 1, 2, or 3.

Exclusion Criteria:

* Patients with concurrent or recent medical conditions that might interfere with study participation, including history of hepatitis, alcohol/substance abuse, uncontrolled psychiatric disorders, known allergy, or contraindication to amide-type local anesthetics, opioids, or propofol.
* Patients who are participating in another study involving an investigational medication within the prior 30 days, or were taking analgesics (ie, non- steroidal anti-inflammatory drugs, acetaminophen, or opioids), antidepressants, or glucocorticoids within the 3 days before surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Score on Numeric Pain Rating Scale | Up to 7 days post-surgery
  A Numeric pain rating scale will be given to the patient on post-operative day (POD) # 1 before discharge and during follow up on POD # 7, and they will be telephoned on subsequent days from discharge till POD # 3 at regular intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil Pappou, MD, PhD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: Undecided
To be decided